

Statistical Analysis Plan

# **Title Page**

Protocol Title: A Phase IV, Multi-center, Open-label, Single-arm 24-hour Ambulatory Blood Pressure Monitoring (ABPM) Study of 16 Weeks Treatment with Androderm® in Hypogonadal Men

**Protocol Number: 3146-402-016** 

**Compound Number: AGN-195263** 

Brief Protocol Title: Androderm® ABPM Study in Hypogonadal Men

**Study Phase: IV** 

Sponsor Name: Allergan Sales, LLC

**Legal Registered Address:** 

Allergan Sales LLC 5 Giralda Farms Madison, NJ 07940

**USA** 

Regulatory Agency Identifying Number(s): NDA 020489, IND 034028

**Approval Date: 28 May 2020** 



# Statistical Analysis Plan

# **Table of Contents**

| Title Pa | age | 1 |
|---|---|---|
| Table o | of Contents | 2 |
| List of | Tables | 3 |
| SAP V | ersion History | 4 |
| 1. | Introduction | 5 |
| 1.1. | Objectives and Endpoints | |
| 1.2. | Study Design | 8 |
| 2. | Statistical Hypotheses | 11 |
| 3. | Sample Size Determination | 12 |
| 4. | Populations for Analysis | 13 |
| 5. | Statistical Analyses | 14 |
| 5.1. | General Considerations | 14 |
| 5.2. | Participant Disposition | 14 |
| 5.3. | Primary Endpoint Analysis | 14 |
| 5.3.1. | Definition of Endpoint | 14 |
| 5.3.2. | Primary Efficacy Analysis | 14 |
| 5.3.3. | Sensitivity Analysis | 14 |
| 5.4. | Secondary and Other Endpoints Analyses | 14 |
| 5.5. | Other Safety Analyses | 16 |
| 5.5.1. | Extent of Exposure. | 16 |
| 5.5.2. | Treatment Compliance | 16 |
| 5.5.3. | Adverse Events | 16 |
| 5. | .5.3.1. Adverse Events of Special Interest | 17 |
| 5.5.4. | Additional Safety Assessments | 17 |
| 5. | .5.4.1. Clinical Laboratory Parameters | 17 |
| 5. | .5.4.2. Vital Signs | 18 |
| 5.6. | Other Analyses | 18 |
| 5.6.1. | Other variables and/or parameters. | 18 |
| 5.6.2. | Subgroup analyses | 18 |
| 5.7. | Interim Analyses | 19 |
| 6. | Supporting Documentation | 20 |
| 6.1. | Appendix 1 List of Abbreviations | 20 |
| 6.2. | Appendix 2: Changes to Protocol-Planned Analyses | 22 |
| 6.3. | Appendix 3: Supporting Study Information | 22 |
| 6.3.1. | Demographics | 22 |
| 6.3.2. | Baseline and Disease Characteristics | 22 |
| 6.3.3. | Protocol Deviations | |
| 6.3.4. | Medical and Surgical History | 22 |
| 6.3.5. | Prior/Concomitant/Follow-up medications (including dictionary) | 22 |



| Androderm | (testosterone transdermal system) | Statistical Analysis Plan |
|---|---|---|
| | verse Events of Special Interest | 23 |
| | tentially Clinically Significant Criteria for Safety Endpoints | |
| 6.3.7.1 | | |
| 0.0.771 | Parameters | |
| 6.3.7.2 | | |
| 6.4. Da | ta handling convention | |
| | alysis Window | |
| 6.4.2. De | rived Efficacy and Health Outcome Data | 26 |
| 6.4.2.1 | . Derivation of Efficacy Endpoints | 26 |
| | peated or Unscheduled Assessments of Safety Parameters | |
| 6.4.4. Mi | ssing Date of the Last Dose of Study treatment | 27 |
| | ssing Severity Assessment for Adverse Events | 27 |
| | ssing Causal Relationship to Study treatment for Adverse | |
| | ents | |
| | ssing Date Imputation | |
| | ssing Date Information for Prior or Concomitant Medication | |
| 6.4.8.1 | F | |
| 6.4.8.2 | F F | |
| 6.4.9. Ch | aracter Values of Clinical Laboratory Parameters | 30 |
| 7. Re | ferences | 31 |
| | List of Tables | |
| Table 1-1 | | 6 |
| Table 1-2 | Schedule of Visits and Procedures | 9 |
| Table 6-1 | Visit Time Windows for Safety Analysis | 25 |
| | List of Figures | |
| Figure 1-1 | Study Design | 8 |



Statistical Analysis Plan

# **SAP Version History**

| SAP Version History Summary | | |
|---|---|---|
| SAP Approval Change Rationale | | |
| 1 | Not Applicable | Original version |



Statistical Analysis Plan

# 1. Introduction

This Statistical Analysis Plan (SAP) provides a technical and detailed elaboration of the statistical analyses of the efficacy and/or safety data as outlined and specified in the final protocol of 3146-402-016 dated 08 Nov 2019. Specifications of tables, figures and data listings are contained in a separate document.



# 1.1. Objectives and Endpoints

# Table 1-1

| Objective<br>Clinical | | |
|---|---|---|
| Category | Statistical Category | Estimand <sup>1</sup> |
| | e: To determine whether Androd osterone replacement treatment. | erm has a meaningful effect on 24-hour average systolic blood pressure (SBP) as measured by ABPM in |
| Efficacy category 1 | Primary | <ul> <li>Variable: change from baseline in 24-hour average SBP obtained at Week 16</li> <li>Population: modified intent-to-treat (mITT)</li> <li>IES: Hypothetical Strategy <ul> <li>Data after treatment discontinuation are treated as missing</li> </ul> </li> <li>PLS: the difference in the variable means between at baseline and at Week 16</li> <li>Descriptive analysis including two-sided 95% confidence interval</li> </ul> |
| | Sensitivity (Missing in 24-<br>hour average SBP at Week<br>16 under missing at<br>random assumption) | Multiple imputation (MI) for missing data |
| | tive: To determine whether Andr<br>one replacement treatment | oderm has a meaningful effect on 24-hour blood pressure (BP) parameters as measured by ABPM in men |
| Efficacy category 2 | Secondary | <ul> <li>Variable: Change from baseline in 24-hour average diastolic blood pressure (DBP), mean arterial pressure (MAP), pulse pressure and heart rate obtained at Week 16.</li> <li>Population: mITT</li> </ul> |
| Exploratory: To treatment | determine whether Androderm ha | as a meaningful effect on BP parameters as measured by ABPM in men who use testosterone replacement |
| Efficacy category 3 | Other | <ul> <li>Change from baseline in daytime average SBP, DBP, MAP, pulse pressure and heart rate obtained<br/>at Week 16</li> </ul> |



CONFIDENTIAL Statistical Analysis Plan

# $And roderm^{\circledR} \ (test osterone \ transdermal \ system)$

| Objective | |
|---|---|
| Clinical | |
| Category Statistical Category | Estimand <sup>1</sup> |
| | Change from baseline in night-time average SBP, DBP, MAP, pulse pressure and heart rate obtained at Week 16 Change from baseline over time (hourly average) by nominal clock time and time after dose: SBP, DBP, MAP, pulse pressure and heart rate Status (yes/no) of participants with new anti-hypertensive medications Status (yes/no) of participants with dose increases in anti-hypertensive medications Outlier responder for participants meeting SBP ≥ 160 mm Hg for 24-hour average Outlier responder for participants meeting SBP change from baseline ≥ 20 mm Hg for 24-hour average Outlier responder for participants meeting DBP ≥ 100 mm Hg for 24-hour average Outlier responder for participants meeting DBP change from baseline ≥ 15 mm Hg for 24-hour average Status (yes/no) of participants with normalized testosterone concentrations at Week 16 fonce daily Androderm for 16 weeks in hypogonadal men. Variable: Presence of TEAEs Population: Safety Analysis: descriptive Variable: change from baseline in clinical laboratory tests and vital sign Population: Safety Analysis: descriptive Variable: potentially clinically significant in clinical laboratory tests and vital sign Population: Safety Analysis: descriptive |

IES = Intercurrent event(s) strategy; PLS = Population-level summary.

<sup>1</sup> All estimand attributes explicitly identified for primary/secondary and select key estimands only.



Statistical Analysis Plan

# 1.2. Study Design

This is a multi-center, open-label, single-arm study in hypogonadal men to evaluate the effect of once daily Androderm on BP parameters as measured by 24-hour ABPM. It is projected that approximately 40 sites in the United States will enroll approximately 150 participants who will receive at least 1 dose for this study.

The study will consist of a screening period of approximately 3 weeks (21 days), followed by an intervention period of 16 weeks (minimum of 113 + 7 days), for a total study duration of approximately 19 weeks (133 days). All participants who meet the criteria for participation in the study will be administered Androderm at the starting dose of 4 mg/day. On Visit 2, study participants will have morning serum concentrations of testosterone measured. If participants have a serum concentration below 400 ng/dL, the dose of Androderm will be increased to 6 mg/day (one 4 mg/day system and one 2 mg/day system). If the serum concentration is above 930 ng/dL, the dose of Androderm will be decreased to 2 mg/day. All others will remain on 4 mg/day.

Approximately 300 participants will be screened to achieve approximately 150 enrolled participants who will receive at least 1 dose and 120 participants with interpretable 24-hour ABPM data at both baseline and the end of Week 16. Participants who prematurely discontinue from the study will not be replaced but will be followed to obtain the last 24-hour ABPM assessment.

Figure 1-1 Study Design



Statistical Analysis Plan

Androderm® (testosterone transdermal system)

Table 1-2 Schedule of Visits and Procedures

| Procedure | S | creenin<br>Period | g | | Intervention Period/Study Day | | | Notes | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit Name | S1 | S2 | S3 | V1 | V2 | V3/TC | V4 | V5 | V6/EOS/ET | V3 only if dose<br>titration is<br>needed,<br>otherwise TC |
| Visit Windows | Up<br>to<br>Day<br>-21 | At<br>least<br>48<br>hours<br>after<br>S1 | Day<br>-3<br>to -<br>1 | Day<br>1 | Day 14 ± 3 | ~Day<br>21 | Day 56 ± 3 | EOS<br>-1 | Day 113 + 7 | V3/TC after V2<br>morning<br>testosterone<br>results are<br>available |
| Informed consent | X | | | | | | | | | |
| Inclusion and exclusion criteria | X | X | X | X | | | | | | Recheck<br>eligibility at V1<br>before dispensing<br>study<br>intervention |
| Demography | X | | | | | | | | | |
| Medical and<br>surgical history<br>(includes prior<br>medications) | X | | | | | | | | | |
| Height and weight | X | | | | | | | | X | Height at S1 only |
| Vital signs | X | X | X | X | X | | X | X | X | Triplicate sitting<br>BP and heart<br>rate; temperature |
| Physical examination | | X | | X | | | | | X | |
| Fasting morning testosterone | х | X | Х | | х | | X | X | | Between 0700<br>and 1100 local<br>time<br>Obtain a fasting<br>morning<br>testosterone<br>sample before<br>ABPM device<br>placement |
| Fasting laboratory assessments | X | | | | | | | | X | Hematology<br>(including PT<br>and INR),<br>chemistry<br>(including liver<br>chemistry and<br>HbA1c), PSA,<br>urinalysis |



# Statistical Analysis Plan

Androderm® (testosterone transdermal system)

| Procedure | S | creenin<br>Period | g | Intervention Period/Study Day | | | | Notes | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit Name | S1 | S2 | S3 | V1 | V2 | V3/TC | V4 | V5 | V6/EOS/ET | V3 only if dose<br>titration is<br>needed,<br>otherwise TC |
| Visit Windows | Up<br>to<br>Day<br>-21 | At<br>least<br>48<br>hours<br>after<br>S1 | Day<br>-3<br>to -<br>1 | Day<br>1 | Day 14 ± 3 | ~Day<br>21 | Day 56 ± 3 | EOS<br>-1 | Day 113 + 7 | V3/TC after V2<br>morning<br>testosterone<br>results are<br>available |
| I-PSS | | X | | | | | | | X | |
| Prostate digital rectal exam | | X | | | | | | | X | Not required if<br>normal digital<br>rectal exam<br>within 6 months<br>of S1; at<br>V6/EOS/ET only<br>if clinically<br>indicated |
| Apply ABPM | | | X | | | | | X | | 24-hour ABPM<br>at ET if feasible |
| Remove ABPM | | | | X | | | | | Х | 24 hours after<br>applying ABPM<br>device |
| Dispense/Begin study intervention | | | | X | | X | | | | At V3 only if<br>dose titration is<br>needed |
| Return/Reconcile study intervention | | | | | | X | | | X | At V3 only if<br>dose titration is<br>needed |
| AE review | ←======→ | | | | | | | | | |
| SAE review | ←=====→ | | | | | | | | | |
| Concomitant medication review | ← | | | | | | | | | |



Statistical Analysis Plan

# 2. Statistical Hypotheses

The null and alternative hypotheses for change from baseline in 24-hour average SBP obtained at baseline and Week 16 (Week 16 minus baseline) are as follows:

 $H_0{:}\ mE$  -  $mB \ge 3.0\ versus\ H_a{:}\ mE$  - mB < 3.0

Where mB and mE are mean 24-hour average SBP obtained at baseline and Week 16 respectively.



Statistical Analysis Plan

# 3. Sample Size Determination

Based on the FDA advice letter dated 24 May 2019, and the assumption that the mean difference in 24-hour SBP obtained at baseline and Week 16 is 0.0, with the upper bound of 3.0 mm Hg and the standard deviation of 10.0 mm Hg, 120 participants with available ABPM data at Week 16 will be required to provide 90% power to reject the null hypothesis at the 2 sided 5% significance level. Assuming a 25% dropout rate, 150 participants will be enrolled.

Approximately 300 participants will be screened, to achieve 150 enrolled who receive ≥ 1 administration of study intervention, for an estimated total of 120 evaluable participants.



Statistical Analysis Plan

# 4. Populations for Analysis

The analysis populations will consist of participants as defined below:

- The mITT population includes all participants with valid baseline ABPM session, who received ≥ 1 administration of study intervention, ≥ 1 post-treatment assessments of SBP, and at least 85% compliance to study intervention for the duration of the study.
- The safety population includes all treated participants who receive ≥ 1 administration of study intervention.



Statistical Analysis Plan

# 5. Statistical Analyses

### **5.1.** General Considerations

The ABPM analyses will be based on the mITT population. Baseline is defined as the last nonmissing assessment before the first application of study intervention. All statistical tests will be 2-sided hypothesis tests performed at the 5% level of significance for main effects. All CIs will be 2-sided 95% CIs, unless stated otherwise. No multiple comparison procedures will be applied.

# 5.2. Participant Disposition

Number of participants screened for the study will be provided.

The summary of study disposition in the Safety population will be provided as treated for the following:

- Number and percentage of participants treated
- Number and percentage of participants completed
- Number and percentage of participants discontinued
- Reasons for discontinuation from study
- In addition, a listing will be provided for participant disposition.

# 5.3. Primary Endpoint Analysis

# **5.3.1.** Definition of Endpoint

The primary efficacy endpoint is change from baseline in 24-hour average SBP obtained at Week 16.

### 5.3.2. Primary Efficacy Analysis

Continuous descriptive statistics (n, mean, SD, median, min, max, Q1 and Q3) of 24-hour average SBP at baseline, Week 16, and change from baseline at Week 16 will be presented. Change from baseline at Week 16 will be tested using paired t-test, along with a 2-sided 95% CI.

If the upper bound of the two-sided 95% CI is less than 3.0, the alternative hypothesis of excluding an increase of 3 mm Hg in SBP will be inferred.

### **5.3.3.** Sensitivity Analysis

Missing value in 24-hour average 24 hours SBP obtained at Week 16 will be imputed using multiple imputation (MI). In the MI analysis, the missing data will be assumed to follow a missing at random (MAR) pattern.

# 5.4. Secondary and Other Endpoints Analyses

Secondary and other efficacy endpoints are defined as follows.



Statistical Analysis Plan

Androderm® (testosterone transdermal system)

Secondary efficacy endpoints:

• Change from baseline in 24-hour average DBP, MAP, pulse pressure, and heart rate obtained at Week 16

#### Other efficacy endpoints:

- Change from baseline in daytime average SBP, DBP, MAP, pulse pressure, and heart rate obtained at Week 16
- Change from baseline in night-time average SBP, DBP, MAP, pulse pressure, and heart rate obtained at Week 16
- Change from baseline over time (hourly average) by nominal clock time and time after dose: SBP, DBP, MAP, pulse pressure, and heart rate
- The status (yes or no) of participants with new anti-hypertensive medications
- The status (yes or no) of participants with dose increases in anti-hypertensive medications
- Outlier responder for participants meeting SBP ≥ 160 mm Hg for 24-hour average and for hourly average
- Outlier responder for participants meeting SBP change from baseline ≥ 20 mm Hg for 24-hour average and for hourly average
- Outlier responder for participants meeting DBP ≥ 100 mm Hg for 24-hour average and for hourly average
- Outlier responder for participants meeting DBP change from baseline ≥ 15 mm Hg for 24-hour average and for hourly average
- Status (yes/no) of participants with normalized testosterone concentrations (within range of 300 to 1030 ng/dL inclusive) at Week 16

Continuous secondary endpoints will be summarized by descriptive statistics (n, mean, SD, median, min, max, Q1 and Q3).

Categorical secondary and other endpoints will be summarized by number and percentage of participants in specified categories.

Plots of hourly average in SBP and DBP included deviation bars for baseline and Week 16.

Cumulative distribution curves of change from baseline in 24-hour average SBP and DBP at Week 16.

Forest plots of daytime, nighttime, and 24-hour change from baseline with 95% confidence interval displays for SBP and DBP.



Statistical Analysis Plan

# 5.5. Other Safety Analyses

# **5.5.1.** Extent of Exposure

The exposure to study intervention, calculated as (*last study intervention date - first study intervention date + I*), will be summarized using descriptive statistics for the Safety population.

Patient-years, defined as exposure to the study intervention in years, will be summarized for the Safety Population

# **5.5.2.** Treatment Compliance

Dosing compliance for a specified period is defined as the number of transdermal systems applied by a patient during that period divided by the number of transdermal systems prescribed for the same period multiplied by 100. This information will be obtained from Study Intervention Record of the patient's electronic case report form.

Descriptive statistics for study intervention compliance will be presented for each period between 2 consecutive visits for the Safety Population.

#### 5.5.3. Adverse Events

Adverse events (AEs) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 22.1 or higher.

An AE will be considered a TEAE if the AE began or worsened (increased in severity or became serious) on or after the date (and time, if known) of the first dose of study intervention. However, an AE that occurs more than 30 days after the last dose of study intervention will not be counted as a TEAE.

An AE will be considered a TESAE if it is a TEAE that additionally meets any SAE criterion.

The number and percentage of participants with TEAEs during the study will be tabulated by system organ class and preferred term and by system organ class, preferred term, and severity.

The number and percentage of participants with treatment-related TEAEs during the study will be tabulated by system organ class and preferred term.

If more than 1 AE is coded to the same preferred term for the same participant, the participant will be counted only once for that preferred term using the most severe and most related occurrence for the summarizations by severity and by relationship to study intervention.

The incidence of common ( $\geq 2\%$  of participants in any treatment group) TEAEs will be summarized by preferred term.

Summary tables will be provided for participants with TESAEs and participants with TEAEs leading to discontinuation if these occurred in 5 or more participants. Listings of all AEs, SAEs, and AEs leading to discontinuation by participant will be presented.



Statistical Analysis Plan

Androderm<sup>®</sup> (testosterone transdermal system)

# **5.5.3.1.** Adverse Events of Special Interest

Potential Hy's Law criteria within a 24-hour window is defined by a post baseline elevation of alanine aminotransferase (ALT) or aspartate aminotransferase (AST)  $\geq$  3 x ULN, along with total bilirubin (TBL)  $\geq$  2 x ULN and a non-elevated alkaline phosphatase (ALP) < 2 x ULN, all based on blood draws collected within a 24-hour period. Potential Hy's Law criteria without time window is defined by maximum of post baseline elevation of ALT or AST  $\geq$  3 x ULN, along with maximum of post baseline elevation of TBL  $\geq$  2 x ULN. Patients who meet the potential Hy's Law criteria from the first dose of study drug to the end of study will be summarized. Supportive tabular displays will also be provided.

Prostate events will be summarized and provided in a listing.

# **5.5.4.** Additional Safety Assessments

For clinical laboratory, vital sign, and ECG, the last nonmissing safety assessment before the first dose of study intervention will be used as the baseline for all analyses of that safety parameter.

### **5.5.4.1.** Clinical Laboratory Parameters

Descriptive statistics for values and changes from the baseline in standard units at each assessment time point will be presented for the following laboratory parameters:

| Laboratory<br>Assessments | Parameters | | | |
|---|---|---|---|---|
| Hematology | Platelet count RBC count Hemoglobin Hematocrit PT INR | RBC indices: MCV MCH MCHC %Reticulocytes | | WBC count with differential (absolute): Neutrophils Lymphocytes Monocytes Eosinophils Basophils |
| Clinical Chemistry | BUN Creatinine Glucose, fasting | Potassium Sodium Calcium | AST ALT Alkaline | Total, direct and indirect bilirubin Total protein Cholesterol, |
| | HbA1c Prolactin | PSA | phosphatas Fasting mo testosterone | e chloride, albumin<br>rning |
| Routine Urinalysis <sup>a</sup> | <ul> <li>Specific gravity</li> <li>pH, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase by dipstick</li> <li>Microscopic examination (if blood or protein is abnormal)</li> </ul> | | | |

Local urine testing will be standard for the protocol unless serum testing is required by local regulation or IRB/IEC.



Statistical Analysis Plan

Androderm® (testosterone transdermal system)

Clinical laboratory test values will be considered potentially clinically significant (PCS) if they meet either the lower-limit or higher-limit PCS criteria listed in Section 6.3.7.1. The number and percentage of participants who have PCS postbaseline clinical laboratory values will be tabulated by study intervention group. The percentages will be calculated relative to the number of participants with available non-PCS baseline values and at least 1 postbaseline assessment for the double-blind treatment period. The numerator will be the total number of participants with available non-PCS baseline values and at least 1 PCS postbaseline value during the study. A supportive tabular display of PCS values will be provided, including the PID number, baseline and all postbaseline values.

In addition, a tabular display showing all AEs that occurred in participants who had PCS postbaseline clinical laboratory values will be provided.

# **5.5.4.2.** Vital Signs

Descriptive statistics for vital signs and their changes from baseline at each assessment timepoint will be presented by study intervention group.

Vital sign values will be considered PCS if they meet both the observed value criterion and the change from baseline value criterion, if both criteria are available, or meet either the observed value criterion or the change from baseline value criterion that will be detailed in Section 6.3.7.2. The number and percentage of participants who have PCS postbaseline vital sign values will be tabulated by study treatment. The percentages will be calculated relative to the number of participants who have available baseline or non-PCS baseline (for parameters with only the observed value criterion) values and at least 1 postbaseline assessment. The numerator will be the total number of participants with at least 1 PCS postbaseline value during the study. A supportive listing of PCS values will be provided. In addition, a tabular display showing all AEs that occurred in participants who had PCS postbaseline vital sign values will be provided.

# 5.6. Other Analyses

### **5.6.1.** Other variables and/or parameters.

#### 5.6.2. Subgroup analyses

Participants without baseline medical history of hypertension, with baseline medical history of hypertension untreated and with baseline medical history of hypertension treated will be performed for following endpoints and graphs.

- Change from baseline in 24-hour average SBP and DSP obtained at Week 16
- Change from baseline hourly average by nominal clock time and time after dose: SBP and DBP
- Outlier responder for participants meeting SBP ≥ 160 mm Hg for 24-hour average and for hourly average



Statistical Analysis Plan

Androderm<sup>®</sup> (testosterone transdermal system)

- Outlier responder for participants meeting SBP change from baseline ≥ 20 mm Hg for 24-hour average and for hourly average
- Outlier responder for participants meeting DBP  $\geq$  100 mm Hg for 24-hour average and for hourly average
- Outlier responder for participants meeting DBP change from baseline ≥ 15 mm Hg for 24-hour average and for hourly average
- Plots of hourly average in SBP and DBP included deviation bars for baseline and Week 16
- Cumulative distribution curves of change from baseline in 24-hour average SBP and DBP at Week 16
- Forest plots of daytime, nighttime, and 24-hour change from baseline with 95% confidence interval displays for SBP and DBP.

# 5.7. Interim Analyses

No interim analysis is planned.



# 6. Supporting Documentation

# **6.1.** Appendix 1 List of Abbreviations

| Abbreviation | Definition |
|---|---|
| ABPM | ambulatory blood pressure monitoring |
| AE | adverse event |
| AESI | adverse event of special interest |
| ALT | alanine aminotransferase |
| AST | aspartate aminotransferase |
| BMI | body mass index |
| BP | blood pressure |
| BUN | blood urea nitrogen |
| CDISC | Clinical Data Interchange Standards Consortium |
| CFR | Code of Federal Regulations |
| CI | confidence interval |
| CIOMS | Council for International Organizations of Medical Sciences |
| CONSORT | Consolidated Standards of Reporting Trials |
| CRF | case report form |
| DBP | diastolic blood pressure |
| DHEA | dehydroepiandrosterone |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EOS | end of study |
| ET | early termination |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| HbA1c | hemoglobin A1c |
| ICF | informed consent form |
| ICH | International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use |
| ID | identification |
| IEC | Independent Ethics Committee |
| INR | international normalized ratio |
| I-PSS | International Prostate Symptom Score |
| IRB | Internal Review Board |
| ISO | International Organization for Standardization |
| IUD | intrauterine device |
| IUS | intrauterine system |



# Statistical Analysis Plan

CONFIDENTIAL Androderm® (testosterone transdermal system)

| Abbreviation | Definition |
|--------------|-----------------------------------------------|
| MAR | missing at random |
| MAP | mean arterial pressure |
| MCH | mean corpuscular hemoglobin |
| MCHC | mean corpuscular hemoglobin concentration |
| MCV | mean corpuscular volume |
| MI | multiple imputation |
| mITT | modified intent-to-treat |
| N/A | not applicable |
| NCI | National Cancer Institute |
| PCS | potentially clinically significant |
| PK | pharmacokinetic |
| PSA | prostate specific antigen |
| PT | prothrombin time |
| Q1 | quartile 1 |
| Q3 | quartile 3 |
| RBC | red blood cell |
| S1 | Screening Visit 1 |
| S2 | Screening Visit 2 |
| S3 | Screening Visit 3 |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SBP | systolic blood pressure |
| SD | standard deviation |
| SoA | schedule of activities |
| SUSAR | suspected unexpected serious adverse reaction |
| TC | teleconference |
| TEAE | treatment-emergent adverse event |
| TESAE | treatment-emergent serious adverse event |
| ULN | upper limit of normal |
| V1 | Intervention Period Visit 1 |
| V2 | Intervention Period Visit 2 |
| V3 | Intervention Period Visit 3 |
| V4 | Intervention Period Visit 4 |
| V5 | Intervention Period Visit 5 |
| V6 | Intervention Period Visit 6 |
| WBC | white blood cell |



CONFIDENTIAL Statistical Analysis Plan Androderm® (testosterone transdermal system)

# 6.2. Appendix 2: Changes to Protocol-Planned Analyses

There are no changes from the protocol-planned analyses.

# 6.3. Appendix 3: Supporting Study Information

# 6.3.1. Demographics

Demographic parameters (eg, age, race, ethnicity, sex) will be summarized descriptively for the Safety Population.

#### 6.3.2. Baseline and Disease Characteristics

Baseline characteristics (weight; height; and body mass index, calculated as weight [kg]/(height [m])2 and baseline medical history of without hypertension, with hypertension untreated and treated will be summarized descriptively for the Safety Population.

#### **6.3.3.** Protocol Deviations

Protocol deviations will be defined in Protocol Deviation Requirement Specification, including importance classification. The number and percentage of participants with important protocol deviations will be summarized for Safety Population.

# **6.3.4.** Medical and Surgical History

Abnormalities in participants' medical and surgical history will be coded using the Medical Dictionary for Regulatory Activities, version 22.1 or higher. The number and percentage of participants with abnormalities in medical and surgical histories in each system organ class and preferred term will be summarized for the Safety Population.

# 6.3.5. Prior/Concomitant/Follow-up medications (including dictionary)

The medication data will be coded using the World Health Organization (WHO) Drug Global B3 version March 2019 or higher.

Prior medication is defined as any medication taken before the first dose of study intervention. Concomitant medication is defined as any medication taken on or after the date of the first dose of study intervention.

The number and percentage of participants reporting prior or concomitant medications will be summarized for ATC class and code, and preferred drug name. If more than one medication is coded to the same preferred drug name for the same participant, the participant will be counted only once for that preferred drug name. Prior and concomitant medications will be summarized separately.



Statistical Analysis Plan

Androderm® (testosterone transdermal system)

# **6.3.6.** Adverse Events of Special Interest

- 1. Potential Hy's Law cases:
  - ALT or AST  $\geq$  3 × ULN and
  - Total Bilirubin  $\geq 2 \times ULN$  and
  - Alkaline Phosphatase < 2 × ULN

Anytime from the time the participant signs the ICF for the trial, until the final follow-up visit, investigators will notify the sponsor immediately when all the above criteria have been met. A potential Hy's law case will be sent directly to the sponsor by emailing

IR-clinical-SAE@allergan.com on an AE of Special Interest Form along with the SAE Report Form as soon as possible (within 24 hours of learning of the potential Hy's Law). The CRF for potential Hy's law cases will be completed within 7 calendar days. Every effort to determine the cause of the liver enzyme abnormalities will be made, and close monitoring will be initiated in conjunction with the medical monitor and in accordance with the FDA "Guidance for Industry: Drug-Induced Liver Injury: Premarketing Clinical Evaluation" July 2009.

#### 2. Prostate events:

• Lower urinary tract symptoms of prostatic hyperplasia

Potential lower urinary tract symptoms of prostatic hyperplasia will be sent directly to the sponsor by emailing IR-clinical-SAE@allergan.com on an AE of Special Interest Form along with the SAE Report Form as soon as possible (within 24 hours of learning of the event). The CRF for lower urinary tract symptoms of prostatic hyperplasia will be completed within 7 calendar days.

### 6.3.7. Potentially Clinically Significant Criteria for Safety Endpoints

The potentially clinically significant criteria for clinical laboratory parameters and vital signs are provided in the following sections.

6.3.7.1. Potential Clinically Significant for Clinical Laboratory Parameters

| Parameter | SI Unit | Lower Limit | Higher Limit |
|---|---|---|---|
| CHEMISTRY | | | |
| Albumin | g/L | < 0.9 × LLN | > 1.1 × ULN |
| Alanine<br>aminotransferase<br>(ALT) | U/L | _ | $\geq$ 3 × ULN |
| Alkaline phosphatase | U/L | _ | ≥ 3 × ULN |



Statistical Analysis Plan

| Parameter | SI Unit | Lower Limit | Higher Limit |
|---|---|---|---|
| Aspartate<br>aminotransferase<br>(AST) | U/L | _ | $\geq$ 3 × ULN |
| Bilirubin, total | μmol/L | _ | > 1.5 × ULN |
| Calcium | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| Chloride | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| Cholesterol, Total | mmol/L | _ | > 1.3× ULN |
| Creatinine | μmol/L | _ | > 1.3 × ULN |
| Glucose, fasting, serum | mmol/L | < 0.8 × LLN | > 1.2× ULN |
| Glucose, random, serum | mmol/L | < 0.8 × LLN | > 1.4 × ULN |
| Potassium | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| Protein, total | g/L | < 0.9 × LLN | > 1.1 × ULN |
| Sodium | mmol/L | < 0.9 × LLN | > 1.1 × ULN |
| Urea Nitrogen (BUN) | mmol/L | _ | > 1.2 × ULN |
| HEMATOLOGY | | | |
| Basophils, absolute cell count | 10 <sup>9</sup> /L | _ | > 3 × ULN |
| Neutrophils, absolute cell count | 10 <sup>9</sup> /L | < 0.8 × LLN | > 1.5 × ULN |
| Hematocrit | Ratio | < 0.9 × LLN | > 1.1 × ULN |
| Hemoglobin | g/L | < 0.9 × LLN | > 1.1 × ULN |
| Platelet count | $10^{9}/L$ | < 0.5 × LLN | > 1.5 × ULN |
| Red blood cell count | $10^{12}/L$ | < 0.9 × LLN | > 1.1 × ULN |
| White blood cell count | 10 <sup>9</sup> /L | < 0.7 × LLN | > 1.5 × ULN |
| URINALYSIS | | | |
| рН | _ | < 0.9 × LLN | > 1.1 × ULN |
| Specific gravity | | | > 1.1 × ULN |

LLN = lower limit of normal value provided by the laboratory; SI = *Le Système International d'Unités* (International System of Units); ULN = upper limit of normal value provided by the laboratory.

Statistical Analysis Plan

6.3.7.2. Potentially Clinically Significant Criteria for Vital Signs

| Parameter | Flag | Criteria | |
|---|---|---|---|
| | | Observed Value | Change from Baseline |
| Systolic blood pressure, mm Hg | High | ≥ 140 | Increase of ≥ 20 |
| | Low | ≤ 90 | Decrease of ≥ 20 |
| Diastolic blood pressure, mm Hg | High | ≥ 90 | Increase of ≥ 15 |
| | Low | ≤ 50 | Decrease of ≥ 15 |
| Pulse rate, bpm | High | ≥ 100 | Increase of ≥ 15 |
| | Low | ≤ 50 | Decrease of ≥ 15 |
| Weight, kg | High | _ | Increase of ≥ 5% |
| | Low | _ | Decrease of ≥ 5% |

SBP = Systolic blood pressure, DBP = Diastolic blood pressure, bpm = beats per minute.

# 6.4. Data handling convention

# 6.4.1. Analysis Window

Table 6-1 presents the visits assigned for analyses and the corresponding range of treatment days (window) during which an actual visit may occur.

Table 6-1 Visit Time Windows for Safety Analysis

| Derived Visit | Scheduled Test / Visit Day <sup>a</sup> | Window |
|---|---|---|
| Day 1 | Day 1 | Days ≤ 1 |
| Week 2 | Day 14 | Days [2, 17] |
| Week 3 | Day 21 | Days [18, 38] |
| Week 8 | Day 56 | Days [39, 79] |
| Week 16 | Day 112 | Days > 79 |
| End of Treatment Period | Final or termination visit du | Final or termination visit during the Treatment Period |



Statistical Analysis Plan

Androderm<sup>®</sup> (testosterone transdermal system)

Test/Visit Day will be calculated as follows: test/visit date – date of the first dose of study drug + 1.

If a participant has 2 or more visits within the same window, the last visit with a nonmissing value will be used for analysis

### 6.4.2. Derived Efficacy and Health Outcome Data

### **6.4.2.1.** Derivation of Efficacy Endpoints

BP parameters, including SBP, DBP, MAP, pulse pressure, and heart rate will be collected by 24-hour ABPM at Baseline and Week 16.

| Term | Definition |
|---|---|
| Baseline ABPM | Any assessment recorded during the approximately 24-hour period starting on Screening Visit 3; after the ABPM device is applied, through Visit 1, when the ABPM device is removed |
| Week 16 (End of study intervention) | Any assessment recorded during the approximately 24-hour period starting on Visit 5, after the ABPM device is applied, through Visit 6/EOS/ET, when the ABPM device is removed |
| 24-hour ABPM | Any assessment recorded at the specified analysis timepoint (baseline, Week 16) during the approximately 24-hour period after the ABPM device is applied through when the ABPM device is removed |
| Daytime ABPM | Any assessment recorded between 0900 and 2100 on either: |
| | the day the ABPM device is applied |
| | the day the ABPM device is removed |
| Night-time ABPM | Any assessment recorded between 0100 and 0600 on either: |
| | the day the ABPM device is applied |
| | the day the ABPM device is removed |
| Hours 0 through 23 | For each Hour X, any assessment recorded between XX00 and XX59, on either: |
| | the day the ABPM device is applied |
| | the day the ABPM device is removed |

Continuous BP endpoints are 24-hour, daytime or night-time average on nonmissing values in BP for baseline, Week 16 or change from baseline at Week 16.

#### 6.4.3. Repeated or Unscheduled Assessments of Safety Parameters

Baseline is defined as the last assessment made before the first dose of study intervention. If endof-study assessments are repeated or if unscheduled visits occur, the last nonmissing postbaseline assessment will be used as the end-of-study assessment for generating summary statistics. However, all postbaseline assessments will be used for PCS value determinations, and all assessments will be presented in the data listings.



Statistical Analysis Plan

Androderm® (testosterone transdermal system)

# 6.4.4. Missing Date of the Last Dose of Study treatment

When the date of the last dose of study intervention is missing, all efforts should be made to obtain the date from the Investigator. If it is still missing after all efforts have been made, the last available study medication date will be used in the calculation of treatment duration.

# 6.4.5. Missing Severity Assessment for Adverse Events

If severity is missing for an AE that started before the date of the first dose of study intervention, an intensity of mild will be assigned. If severity is missing for an AE that started on or after the date of the first dose of study intervention, an intensity of severe will be assigned. The imputed values for severity assessment will be used for the incidence summary; the values will be shown as missing in the data listings.

# 6.4.6. Missing Causal Relationship to Study treatment for Adverse Events

If the causal relationship to the study intervention is missing for an AE that started on or after the date of the first dose of study intervention, a causality of yes will be assigned. The imputed values for causal relationship to double-blind treatment will be used for the incidence summary; the values will be shown as missing in the data listings.

# **6.4.7.** Missing Date Imputation

The following imputation rules only apply to cases in which the start date for AEs is incomplete (ie, partly missing).

#### Missing month and day

If the year of the incomplete start date is the same as the year of the first dose of study intervention, the month and day of the first dose of study intervention will be assigned to the missing fields

If the year of the incomplete start date is before the year of the first dose of study intervention, December 31 will be assigned to the missing fields

If the year of the incomplete start date is after the year of the first dose of study intervention, *January 1* will be assigned to the missing fields

### Missing month only

If only the month is missing, the day will be treated as missing and both the month and the day will be replaced according to the above procedure

#### Missing day only

If the month and year of the incomplete start date are the same as the month and year of the first dose of study intervention, the day of the first dose of study intervention will be assigned to the missing day



Statistical Analysis Plan

Androderm® (testosterone transdermal system)

If either the year of the incomplete start date is before the year of the date of the first dose of study intervention or if both years are the same but the month of the incomplete start date is before the month of the date of the first dose of study intervention, the last day of the month will be assigned to the missing day

If either the year of the incomplete start date is after the year of the date of the first dose of study intervention or if both years are the same but the month of the incomplete start date is after the month of the date of the first dose of study intervention, the first day of the month will be assigned to the missing day

If the stop date is complete and the imputed start date as above is after the stop date, the start date will be imputed by the stop date.

If the start date is completely missing and the stop date is complete, the following algorithm will be used to impute the start date:

• If the stop date is after the date of the first dose of study intervention, the date of the first dose of study intervention will be assigned to the missing start date

If the stop date is before the date of the first dose of study intervention, the stop date will be assigned to the missing start date

# 6.4.8. Missing Date Information for Prior or Concomitant Medications

For prior or concomitant medications, including rescue medications, incomplete (ie, partly missing) start dates and/or stop dates will be imputed. When the start date and the stop date are both incomplete for a participant, the start date will be imputed first.

# **6.4.8.1.** Incomplete Start Date

The following rules will be applied to impute the missing numeric fields for an incomplete prior or concomitant medication start date. If the stop date is complete (or imputed) and the imputed start date is after the stop date, the start date will be imputed using the stop date.

### Missing month and day

If the year of the incomplete start date is the same as the year of the first dose of study intervention, the month and day of the first dose of study intervention will be assigned to the missing fields

If the year of the incomplete start date is before the year of the first dose of study intervention, December 31 will be assigned to the missing fields

If the year of the incomplete start date is after the year of the first dose of study intervention, January 1 will be assigned to the missing fields

# Missing month only

If only the month is missing, the day will be treated as missing and both the month and the day will be replaced according to the above procedure



Statistical Analysis Plan

# Missing day only

If the month and year of the incomplete start date are the same as the month and year of the first dose of study intervention, the day of the first dose of study intervention will be assigned to the missing day

If either the year of the incomplete start date is before the year of the date of the first dose of study intervention or if both years are the same but the month of the incomplete start date is before the month of the date of the first dose of study intervention, the last day of the month will be assigned to the missing day.

If either the year of the incomplete start date is after the year of the date of the first dose of study intervention or if both years are the same but the month of the incomplete start date is after the month of the date of the first dose of study intervention, the first day of the month will be assigned to the missing day

# **6.4.8.2. Incomplete Stop Date**

The following rules will be applied to impute the missing numeric fields for an incomplete prior or concomitant medication stop date. If the date of the last dose of study treatment is missing, replace it with the last visit date in the imputations described below. If the imputed stop date is before the start date (imputed or nonimputed start date), the imputed stop date will be equal to the start date

# Missing month and day

If the year of the incomplete stop date is the same as the year of the last dose of study treatment, the month and day of the last dose of study treatment will be assigned to the missing fields

If the year of the incomplete stop date is before the year of the last dose of study treatment, December 31 will be assigned to the missing fields

If the year of the incomplete stop date is after the year of the last dose of study treatment, January 1 will be assigned to the missing fields

# Missing month only

If only the month is missing, the day will be treated as missing and both the month and the day will be replaced according to the above procedure

#### Missing day only

If the month and year of the incomplete stop date are the same as the month and year of the last dose of study treatment, the day of the last dose of study treatment will be assigned to the missing day

If either the year of the incomplete stop date is before the year of the date of the last dose of study treatment or if both years are the same but the month of the incomplete stop date is before the month of the date of the last dose of study treatment, the last day of the month will be assigned to the missing day



Statistical Analysis Plan

Androderm® (testosterone transdermal system)

If either the year of the incomplete stop date is after the year of the date of the last dose of study treatment or if both years are the same but the month of the incomplete stop date is after the month of the date of the last dose of study treatment, the first day of the month will be assigned to the missing day

# 6.4.9. Character Values of Clinical Laboratory Parameters

If the reported value of a clinical laboratory parameter cannot be used in a statistical summary table because, for example, a character string is reported for a parameter of the numeric type, a coded value must be appropriately determined for use in the statistical analyses. The actual values, however, as reported in the database will be presented in the data listings.



Statistical Analysis Plan

# 7. References

None.